CLINICAL TRIAL: NCT06622967
Title: Multinational Clinical Trial of Real-time Artificial Intelligence System (CadAI-B) for Breast Ultrasound: Prospective Clinical Validation Study
Brief Title: KNUCH CadAI-B-1(KCB-1)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JeeYeon Lee (Other)
Collaborators: Kyungpook National University Chilgok Hospital (Other); BeamWorks Inc. (Industry)
Responsible Party: Sponsor-Investigator, JeeYeon Lee, Associate professor, Kyungpook National University Chilgok Hospital
Organization: Kyungpook National University Chilgok Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KNUCH IRB number : 2024-05-026; Digital healthcare demonstrati (Other: Daegu Gyeongbuk Medical Innovation Foundation)
Record Dates: First submitted 2024-09-17; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Breast Neoplasm; Female
Keywords: breast neoplasm; ultrasound
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CadAI-B intervention group (Experimental): Participants in this arm will receive the CadAI-B system for the detection of lesions. The AI-based tool will assist healthcare professionals in identifying lesions through enhanced image analysis.
  Interventions: Diagnostic Test: CadAI-B

INTERVENTIONS:
Diagnostic Test: CadAI-B — The ultrasound is performed following the usual process. If there are any lesions or areas of concern identified by the patient, a more detailed analysis is conducted on the affected area.
  When a lesion is confirmed, the examiner verifies the results through the frozen image, while also securing the results displayed on CadAI-B.
  The examiner uses the analysis from CadAI-B as a reference to make the final BI-RADS classification.
  Static images and cine clips are captured from the most suspicious areas.

SUMMARY:
The CadAI-B (Computer Aided Design Artificial Intelligence-Breast) system is a real-time AI diagnostic tool for breast ultrasound. It integrates with ultrasound devices to detect suspicious lesions, providing size, BI-RADS, and malignancy probability. After installation and user training, the system displays real-time breast conditions and automatically analyzes lesions when a freeze frame is set, showing results in seconds. This study will assess CadAI-B's accuracy and reliability by comparing its findings with biopsy results.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 years or older
* Individuals scheduled to undergo breast ultrasound for diagnostic evaluation
* Patients whose Ground Truth can be determined through biopsy, surgery, or follow-up

Exclusion Criteria:

* Images containing artifacts that may affect the interpretation
* Presence of breast implants
* Significant breast trauma or mastitis at the time of the breast ultrasound that could cause distortion in image interpretation
* History of surgery or chemotherapy

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female
Enrollment: 100 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Lesion and Per-patient Diagnostic Performance | At the end of the trial, up to 6 months
  AUC (Area Under the Curve), Sensitivity, Specificity

SECONDARY OUTCOMES:
Lesion and Per-patient Detection Performance | At the end of the trial, up to 6 months
  Sensitivity, Specificity

OTHER OUTCOMES:
BeamWorks Usability Evaluation Scale (Score of BeamWorks System Usability Scale (SUS)) | At the end of the trial, up to 6 months
  12~30 : Unacceptable, 30~40 :Marginal, >40:Acceptable

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyeon Lee, MD, PhD, Study Chair — Kyungpook National University Chilgok Hospital
Locations (1):
- Kyungpook National University Chilgok Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No